CLINICAL TRIAL: NCT06144125
Title: Prothrombin Complex Concentrate and Fresh Frozen Plasma in Viscoelastic Test-based Goal-directed Bleeding Management in Cardiac Surgery
Brief Title: Prothrombin Complex Concentrate vs Fresh Frozen Plasma in Goal-directed Bleeding Management in Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC22195220002004
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Valve Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: Patients are randomly divided into two groups (experimental vs control groups).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fresh frozen plasma (Active Comparator): according to the Rotational thromboelastometry (ROTEM) test, CT-EXTEM prolongation, fresh frozen plasma transfusion (FFP) is performed
  Interventions: Biological: fresh frozen plasma
- prothrombin complex concentrate (Experimental): according to the Rotational thromboelastometry (ROTEM) test, CT-EXTEM prolongation, prothrombin complex concentrate (PCC) is administered
  Interventions: Biological: prothrombin complex concentrate

INTERVENTIONS:
Biological: fresh frozen plasma — transfusion of fresh frozen plasma
  Arms: fresh frozen plasma
Biological: prothrombin complex concentrate — prothrombin complex concentrate administration
  Arms: prothrombin complex concentrate

SUMMARY:
The primary endpoint of this study is the completion time of hemostasis treatment when administered Fresh frozen plasma (FFP) and frozen powder coagulation factor concentrate (PCC) in goal-directed bleeding management for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery

Exclusion Criteria:

* thrombocytopenia
* oral anti-coagulant
* anti platelet agents

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
treatment time | 1 min
  duration from the time diagnosing CT-EXTEM prolongation to the time achieving bleeding control

SECONDARY OUTCOMES:
Red Blood Cell amount | I hour
  Red Blood Cell transfusion amount during surgery
FFP amount | 1 hour
  Red Blood Cell transfusion amount during surgery
Platelet amount | 1 hour
  Platelet transfusion amount during surgery
CT-EXTEM | 10 min
  clotting time-EXTEM after PCC or FFP
MA-EXTEM | 10 min
  Maximal amplitude-EXTEM after PCC or FFP
MA-FIBTEM | 10 min
  Maximal amplitude-FIBTEM after PCC or FFP
Postoperative bleeding | 24 hour
  chest tube drainage at postoperative 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD PhD, Principal Investigator — Konkuk University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided